CLINICAL TRIAL: NCT01641770
Title: Oral Nutritional Supplementation in Hospital Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK83
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary Counseling + ONS (Experimental)
  Interventions: Other: Nutritional beverage 10003RF; Other: Dietary Counseling
- Dietary Counseling (Active Comparator)
  Interventions: Other: Dietary Counseling

INTERVENTIONS:
Other: Nutritional beverage 10003RF — 2 sachets per day
  Arms: Dietary Counseling + ONS
Other: Dietary Counseling — Guidelines for dietary counseling include energy and nutrient requirements.
  Arms: Dietary Counseling + ONS
Other: Dietary Counseling — Guidelines for dietary counseling include energy and nutrient requirements.
  Arms: Dietary Counseling

SUMMARY:
The study objective is to evaluate the benefits of Oral Nutritional Supplementation (ONS) plus Dietary Counseling (DC) in newly admitted hospital subjects with moderate or severe malnutrition.

DETAILED DESCRIPTION:
Approximately 212 subjects (men and women) from multiple Institutions in India will participate in this study. Eligible subjects will be randomized into 2 treatment groups.

* Dietary Counseling only (n=106)
* Dietary Counseling + ONS (n=106)

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Recently admitted into hospital ≤36 hrs.
* Identified as having "moderate malnutrition" or "severe malnutrition".
* Anticipated length of hospital stay of at least 3 days.
* Life expectancy of ≥ 12 weeks
* Able to consume foods and beverages orally.
* Willing to abstain from nutritional supplements throughout the study period unless provided be study.

Exclusion Criteria:

* Alcohol or substance abuse, severe dementia, brain metastases, eating disorders or any psychological condition that may interfere with dietary intake, severe nausea, dysphagia, vomiting, diarrhea, active gastritis, gastrointestinal bleeding or other gastrointestinal disturbances.
* Diabetes, burn injury covering greater than or equal to 15% of the body, advanced renal or hepatic disease, active malignancy.
* Ascites, pleural effusion, severe edema or dehydration.
* Severe edema.
* Medications/ supplements/substances that could profoundly modulate metabolism or weight
* Active tuberculosis, acute Hepatitis B or C, or HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2010-10; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in Body weight | baseline and weeks 4, 8, 12

SECONDARY OUTCOMES:
Nutrition Assessment | baseline and week 12
BMI | baseline and week 12
Blood Chemistries (pre-albumin g/L, alpha-1 acid glycoprotein g/L) | baseline and weeks 4,8,12
  values and changes from baseline
Blood Chemistries (albumin gm/dL, hemoglobin gm/dL, total protein gm/dL) | baseline and weeks 4, 8, 12
  values and changes from baseline
Blood Chemistries (glucose mg/dL, creatinine mg/dL) | Baseline and weeks 4,8,12
  values and changes from baseline
Blood Chemistries (c-reactive protein mg/L) | Baseline and weeks 4,8,12
  Values and changes from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Vinita Satyavrat, MD, Study Chair — Abbott Nutrition International-India
Locations (13):
- India (13):
  - King George Hospital / Andhra Medical College, Andhra Pradesh
  - St. Theresa's Hospital, Andhra Pradesh
  - Care Hospital- Hyderabad, Hyderabad
  - Advanced Medicare and Research Institute, Kolkata
  - Sengupta Hospital & Research Institute, Maharashtra
  - Lokmanya Tilak Muncipal Medical College & Lokmanya Thilak Municipal General Hospital, Mumbai
  - Seth GS Medical College and KEM Hospital, Mumbai
  - TN Medical College & BYL Nair Hospital, Mumbai
  - Abhinav Hospital, Nagpur
  - Sir Ganga Ram Hospital, New Delhi
  - Metro Multispecialty Hospital- X-1,Sector, Noida
  - Jehangir Clinical Development Centre Pvt. Ltd., Jehangir Hospital, Pune
  - Immunology at Dayanand Medical College & Hospital, Punjab